CLINICAL TRIAL: NCT00354003
Title: Impact of Disclosure of Dopamine Transporter Imaging Studies in PD Clinical Trials
Brief Title: The Study of the Impact of Disclosing Imaging Study Information to Trial Participants
Status: Completed | Type: Observational
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Other Study IDs: IMAG-DIS 01
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Parkinsonian Syndrome; Parkinson
Keywords: Parkinson; Imaging
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: A series of questionnaires — Research participants who previously underwent ß-CIT imaging will be contacted by the staff at IND to enquire whether they would like to receive their ß-CIT scan data. After signing a Research Participant Information and Consent Form, all research participants will be asked to complete a questionnaire prior to receipt of their imaging data. Those research participants requesting imaging data will be sent their data by IND and may review their data with IND (by phone) and/ or with their study investigator. All research participants will be asked to respond to a second questionnaire after receiving their imaging data and to a third study questionnaire approximately six weeks following receipt of their imaging data.

SUMMARY:
The overall goal of the study is to evaluate how research participants in Parkinson Disease studies that include brain imaging with a dopamine transporter ligand choose to receive the imaging data and what is the impact of the imaging data information on the management of their symptoms.

DETAILED DESCRIPTION:
Research participants who previously underwent ß-CIT imaging will be contacted by the staff at IND to enquire whether they would like to receive their ß-CIT scan data. After signing a Research Participant Information and Consent Form, all research participants will be asked to complete a questionnaire prior to receipt of their imaging data. Those research participants requesting imaging data will be sent their data by IND and may review their data with IND (by phone) and/ or with their study investigator. All research participants will be asked to respond to a second questionnaire after receiving their imaging data and to a third study questionnaire approximately six weeks following receipt of their imaging data.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in imaging study as described within the protocol

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Research participants who previously underwent ß-CIT imaging
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-06-27 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Marek, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Asenbaum S, Brucke T, Pirker W, Podreka I, Angelberger P, Wenger S, Wober C, Muller C, Deecke L. Imaging of dopamine transporters with iodine-123-beta-CIT and SPECT in Parkinson's disease. J Nucl Med. 1997 Jan;38(1):1-6. PMID 8998140
- [Background] Mozley PD, Schneider JS, Acton PD, Plossl K, Stern MB, Siderowf A, Leopold NA, Li PY, Alavi A, Kung HF. Binding of [99mTc]TRODAT-1 to dopamine transporters in patients with Parkinson's disease and in healthy volunteers. J Nucl Med. 2000 Apr;41(4):584-9. PMID 10768556
- [Background] Booij J, Habraken JB, Bergmans P, Tissingh G, Winogrodzka A, Wolters EC, Janssen AG, Stoof JC, van Royen EA. Imaging of dopamine transporters with iodine-123-FP-CIT SPECT in healthy controls and patients with Parkinson's disease. J Nucl Med. 1998 Nov;39(11):1879-84. PMID 9829575
- [Background] Innis RB, Seibyl JP, Scanley BE, Laruelle M, Abi-Dargham A, Wallace E, Baldwin RM, Zea-Ponce Y, Zoghbi S, Wang S, et al. Single photon emission computed tomographic imaging demonstrates loss of striatal dopamine transporters in Parkinson disease. Proc Natl Acad Sci U S A. 1993 Dec 15;90(24):11965-9. doi: 10.1073/pnas.90.24.11965. PMID 8265656
- [Background] Kaufman MJ, Madras BK. Severe depletion of cocaine recognition sites associated with the dopamine transporter in Parkinson's-diseased striatum. Synapse. 1991 Sep;9(1):43-9. doi: 10.1002/syn.890090107. PMID 1796351
- [Background] Niznik HB, Fogel EF, Fassos FF, Seeman P. The dopamine transporter is absent in parkinsonian putamen and reduced in the caudate nucleus. J Neurochem. 1991 Jan;56(1):192-8. doi: 10.1111/j.1471-4159.1991.tb02580.x. PMID 1987318
- [Background] Wilson JM, Levey AI, Rajput A, Ang L, Guttman M, Shannak K, Niznik HB, Hornykiewicz O, Pifl C, Kish SJ. Differential changes in neurochemical markers of striatal dopamine nerve terminals in idiopathic Parkinson's disease. Neurology. 1996 Sep;47(3):718-26. doi: 10.1212/wnl.47.3.718. PMID 8797470
- [Background] Huang WS, Lin SZ, Lin JC, Wey SP, Ting G, Liu RS. Evaluation of early-stage Parkinson's disease with 99mTc-TRODAT-1 imaging. J Nucl Med. 2001 Sep;42(9):1303-8. PMID 11535717
- [Background] Booij J, Tissingh G, Boer GJ, Speelman JD, Stoof JC, Janssen AG, Wolters EC, van Royen EA. [123I]FP-CIT SPECT shows a pronounced decline of striatal dopamine transporter labelling in early and advanced Parkinson's disease. J Neurol Neurosurg Psychiatry. 1997 Feb;62(2):133-40. doi: 10.1136/jnnp.62.2.133. PMID 9048712
- [Background] Fischman AJ, Bonab AA, Babich JW, Palmer EP, Alpert NM, Elmaleh DR, Callahan RJ, Barrow SA, Graham W, Meltzer PC, Hanson RN, Madras BK. Rapid detection of Parkinson's disease by SPECT with altropane: a selective ligand for dopamine transporters. Synapse. 1998 Jun;29(2):128-41. doi: 10.1002/(SICI)1098-2396(199806)29:23.0.CO;2-9. PMID 9593103
- [Background] Seibyl JP, Marek KL, Quinlan D, Sheff K, Zoghbi S, Zea-Ponce Y, Baldwin RM, Fussell B, Smith EO, Charney DS, van Dyck C, et al. Decreased single-photon emission computed tomographic [123I]beta-CIT striatal uptake correlates with symptom severity in Parkinson's disease. Ann Neurol. 1995 Oct;38(4):589-98. doi: 10.1002/ana.410380407. PMID 7574455
- [Background] Volkow ND, Fowler JS, Wang GJ, Logan J, Schlyer D, MacGregor R, Hitzemann R, Wolf AP. Decreased dopamine transporters with age in health human subjects. Ann Neurol. 1994 Aug;36(2):237-9. doi: 10.1002/ana.410360218. PMID 8053661
- [Background] van Dyck CH, Seibyl JP, Malison RT, Laruelle M, Zoghbi SS, Baldwin RM, Innis RB. Age-related decline in dopamine transporters: analysis of striatal subregions, nonlinear effects, and hemispheric asymmetries. Am J Geriatr Psychiatry. 2002 Jan-Feb;10(1):36-43. PMID 11790633
- [Background] Khan NL, Brooks DJ, Pavese N, Sweeney MG, Wood NW, Lees AJ, Piccini P. Progression of nigrostriatal dysfunction in a parkin kindred: an [18F]dopa PET and clinical study. Brain. 2002 Oct;125(Pt 10):2248-56. doi: 10.1093/brain/awf237. PMID 12244082
- [Background] Dekker M, Bonifati V, van Swieten J, Leenders N, Galjaard RJ, Snijders P, Horstink M, Heutink P, Oostra B, van Duijn C. Clinical features and neuroimaging of PARK7-linked parkinsonism. Mov Disord. 2003 Jul;18(7):751-7. doi: 10.1002/mds.10422. PMID 12815653
- [Background] Mozley PD, Acton PD, Barraclough ED, Plossl K, Gur RC, Alavi A, Mathur A, Saffer J, Kung HF. Effects of age on dopamine transporters in healthy humans. J Nucl Med. 1999 Nov;40(11):1812-7. PMID 10565775
- [Background] Catafau AM, Tolosa E; DaTSCAN Clinically Uncertain Parkinsonian Syndromes Study Group. Impact of dopamine transporter SPECT using 123I-Ioflupane on diagnosis and management of patients with clinically uncertain Parkinsonian syndromes. Mov Disord. 2004 Oct;19(10):1175-82. doi: 10.1002/mds.20112. PMID 15390019
- [Background] Jennings DL, Seibyl JP, Oakes D, Eberly S, Murphy J, Marek K. (123I) beta-CIT and single-photon emission computed tomographic imaging vs clinical evaluation in Parkinsonian syndrome: unmasking an early diagnosis. Arch Neurol. 2004 Aug;61(8):1224-9. doi: 10.1001/archneur.61.8.1224. PMID 15313838
- [Background] Whone, A., et al., The REAL-PET study: Slower progression in early Parkinson's disease treated with ropinirole compared with L-Dopa. Neurology, 2002. 58 (suppl3): p. A82-A83.
- [Background] Parkinson Study Group, Levodopa and the progression of Parkinson disease. NEMJ, 2004. 351: p. 18-28.
- [Background] Marek, K., J. Seibyl, and Parkinson Study Group, ß-CIT Scans without evidence of dopaminergic deficit (SWEDD) in the ELLDOPA-CIT and CALM-CIT study: long-term imaging assessment. Neurology, 2003. 60 (Suppl 1): p. A298.